CLINICAL TRIAL: NCT05586126
Title: AnaConDa-therapy in COVID-19 Patients
Status: Terminated | Type: Observational
Why Stopped: Concerns about possible association between drug and increased ICU mortality
Sponsor: Jeroen Bosch Ziekenhuis (Other)
Responsible Party: Principal Investigator, K.S. Simons, MD, PhD, Jeroen Bosch Ziekenhuis
Other Study IDs: 2020.10.15.03
Record Dates: First submitted 2021-01-15; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: COVID-19; SARS CoV-2
Keywords: sevoflurane; propofol; midazolam; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Sevoflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sevoflurane: patients admitted because of respiratory insufficiency due to COVID-19 with need for invasive mechanical ventilation that are sedated by using sevoflurane
  Interventions: Drug: Sevoflurane
- Control: patients admitted because of respiratory insufficiency due to COVID-19 with need for invasive mechanical ventilation that are sedated by means of intravenous medication, such as propofol, midazolam, esketamine of fentanyl

INTERVENTIONS:
Drug: Sevoflurane — sevoflurane inhalation
  Groups: Sevoflurane

SUMMARY:
COVID 19-pneumonia may evolve into respiratory insufficiency for which invasive mechanical ventilation is required. Recently, inhaled anesthetics have become available for sedation of critically ill patients. Based upon recent research, these anesthetics may provide advantages in improvement of P/F ratio in ARDS patients. However, up to now, its effects on COVID-19 pneumonia patients is unknown; therefore, this study was designed as a plan to investigate whether the use of inhaled sevoflurane leads to improvement of oxygenation compared to intravenous sedatives in mechanically ventilated COVID-19 patients

DETAILED DESCRIPTION:
COVID-19 is an infectious disease caused by the virus SARS-CoV-2, which can lead to severe pneumonia with acute respiratory distress syndrome (ARDS)-like presentation. In this condition, the exchange of oxygen and carbon dioxide in the lungs is compromised because of an inflammatory response with capillary leak. This leads to deterioration of oxygenation with hypoxemia and a decrease in P/F (arterial oxygen tension/fraction of inspired oxygen) ratio, resulting in need for invasive mechanical ventilation. To accomplish this, the patient needs to be sedated. Classic, intravenous sedatives usually come with long half-lifes, which lead to prolonged need for mechanical ventilation, because of residual sedation. Next to short half-life, the inhalation anesthetic sevoflurane is supposed to have anti-inflammatory effects, which could improve oxygenation.

This study is designed to investigate the hypothesis that sedation by use of sevoflurane leads to better oxygenation in COVID-19 patients, compared to intravenous sedatives.

Secondarily, the effects of sevoflurane compared to intravenous sedatives on duration of admission and mechanical ventilation, on respiratory parameters and hemodynamics, inflammatory parameters, use of opioids, manner of waking up and prevalence of delirium, will be investigated.

Study design: The study concerns a single center cohort study in the ICU of the Jeroen Bosch Hospital in The Netherlands. Inhaled anesthesia by sevoflurane is compared to intravenous sedation. Both are considered to be standard of care.

Study population: Patients with respiratory insufficiency due to COVID-19 pneumonia, with need for invasive mechanical ventilation on the ICU in the Jeroen Bosch Hospital.

Study parameters: Primary outcome is P/F ratio (arterial oxygen tension/fraction of inspired oxygen; PaO2/FiO2 ratio) on day 2 and day 5. Secondary outcomes are duration of ICU admission, number of ventilator-free days after 28 days (28VFD), inflammation parameters (CRP/PCT), quality of waking up, number of delirium free days after 28 days (28DFD) and need for vasopressors. Also patient characteristics like demographic information (age, sex, BMI, comorbidity), respiratory and hemodynamic values and use of other sedatives will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* More than 24 hours of invasive mechanical ventilation needed
* Positive test (e.g. Polymerase Chain Reaction (PCR)) for SARS-CoV-2

Exclusion Criteria:

* pulmonary history
* known allergy or hypersensitivity for halogenated anesthetics
* known or suspected predisposition for malignant hyperthermia
* suspected or proven intracranial hypertension
* severe liver dysfunction and/or icterus (serum bilirubin >42,8-51,3 μg per liter)
* neutropenia (<0.5X10^9 neutrophils per liter)
* chemotherapy in the month prior to ICU admission
* patients that are transported to other hospitals during admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with proven COVID-19 and need for invasive mechanical ventilation in the ICU of the Jeroen Bosch Hospital
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
P/F ratio | day 2 after intubation
  arterial oxygen tension divided by fraction of inspired oxygen

SECONDARY OUTCOMES:
duration of ICU admission | through ICU admission
  number of days of admission
28VFD | 28 days after intubation
  number of ventilator-free days after 28 days
28DFD | 28 days after intubation
  number of delirium-free days after 28 days
need for vasopressors | duration of ICU stay
  cumulative dosage per day
28DM | 28 days after intubation
  mortality after 28 days
P/F ratio day 5 | day 5 after intubation
  P/F ratio on day 5 after intubation

CONTACTS AND LOCATIONS:
Overall Officials: D. van Nieuwenhuizen, RN, Principal Investigator — Jeroen Bosch Hospital
Locations (1):
- Jeroen Bosch Ziekenhuis, 's-Hertogenbosch, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Banks WA, Kastin AJ, Gutierrez EG. Penetration of interleukin-6 across the murine blood-brain barrier. Neurosci Lett. 1994 Sep 26;179(1-2):53-6. doi: 10.1016/0304-3940(94)90933-4. PMID 7845624
- [Background] Bernard GR, Artigas A, Brigham KL, Carlet J, Falke K, Hudson L, Lamy M, LeGall JR, Morris A, Spragg R. Report of the American-European consensus conference on ARDS: definitions, mechanisms, relevant outcomes and clinical trial coordination. The Consensus Committee. Intensive Care Med. 1994;20(3):225-32. doi: 10.1007/BF01704707. PMID 8014293
- [Background] Bisbal M, Arnal JM, Passelac A, Sallee M, Demory D, Donati SY, Granier I, Corno G, Durand-Gasselin J. [Efficacy, safety and cost of sedation with sevoflurane in intensive care unit]. Ann Fr Anesth Reanim. 2011 Apr;30(4):335-41. doi: 10.1016/j.annfar.2011.01.019. Epub 2011 Mar 15. French. PMID 21411266
- [Background] Burki T. The origin of SARS-CoV-2. Lancet Infect Dis. 2020 Sep;20(9):1018-1019. doi: 10.1016/S1473-3099(20)30641-1. No abstract available. PMID 32860762
- [Background] Ferrando C, Aguilar G, Piqueras L, Soro M, Moreno J, Belda FJ. Sevoflurane, but not propofol, reduces the lung inflammatory response and improves oxygenation in an acute respiratory distress syndrome model: a randomised laboratory study. Eur J Anaesthesiol. 2013 Aug;30(8):455-63. doi: 10.1097/EJA.0b013e32835f0aa5. PMID 23545542
- [Background] Gattinoni L, Chiumello D, Caironi P, Busana M, Romitti F, Brazzi L, Camporota L. COVID-19 pneumonia: different respiratory treatments for different phenotypes? Intensive Care Med. 2020 Jun;46(6):1099-1102. doi: 10.1007/s00134-020-06033-2. Epub 2020 Apr 14. No abstract available. PMID 32291463
- [Background] Grifoni E, Valoriani A, Cei F, Lamanna R, Gelli AMG, Ciambotti B, Vannucchi V, Moroni F, Pelagatti L, Tarquini R, Landini G, Vanni S, Masotti L. Interleukin-6 as prognosticator in patients with COVID-19. J Infect. 2020 Sep;81(3):452-482. doi: 10.1016/j.jinf.2020.06.008. Epub 2020 Jun 8. No abstract available. PMID 32526326
- [Background] Jabaudon M, Boucher P, Imhoff E, Chabanne R, Faure JS, Roszyk L, Thibault S, Blondonnet R, Clairefond G, Guerin R, Perbet S, Cayot S, Godet T, Pereira B, Sapin V, Bazin JE, Futier E, Constantin JM. Sevoflurane for Sedation in Acute Respiratory Distress Syndrome. A Randomized Controlled Pilot Study. Am J Respir Crit Care Med. 2017 Mar 15;195(6):792-800. doi: 10.1164/rccm.201604-0686OC. PMID 27611637
- [Background] Jerath A, Ferguson ND, Cuthbertson B. Inhalational volatile-based sedation for COVID-19 pneumonia and ARDS. Intensive Care Med. 2020 Aug;46(8):1563-1566. doi: 10.1007/s00134-020-06154-8. Epub 2020 Jun 25. PMID 32588067
- [Background] Jerath A, Parotto M, Wasowicz M, Ferguson ND. Volatile Anesthetics. Is a New Player Emerging in Critical Care Sedation? Am J Respir Crit Care Med. 2016 Jun 1;193(11):1202-12. doi: 10.1164/rccm.201512-2435CP. PMID 27002466
- [Background] Kellner P, Muller M, Piegeler T, Eugster P, Booy C, Schlapfer M, Beck-Schimmer B. Sevoflurane Abolishes Oxygenation Impairment in a Long-Term Rat Model of Acute Lung Injury. Anesth Analg. 2017 Jan;124(1):194-203. doi: 10.1213/ANE.0000000000001530. PMID 27782948
- [Background] Mesnil M, Capdevila X, Bringuier S, Trine PO, Falquet Y, Charbit J, Roustan JP, Chanques G, Jaber S. Long-term sedation in intensive care unit: a randomized comparison between inhaled sevoflurane and intravenous propofol or midazolam. Intensive Care Med. 2011 Jun;37(6):933-41. doi: 10.1007/s00134-011-2187-3. Epub 2011 Mar 29. PMID 21445642
- [Background] O'Gara B, Talmor D. Lung protective properties of the volatile anesthetics. Intensive Care Med. 2016 Sep;42(9):1487-9. doi: 10.1007/s00134-016-4429-x. Epub 2016 Jul 4. No abstract available. PMID 27376746
- [Background] Perbet S, Bourdeaux D, Sautou V, Pereira B, Chabanne R, Constantin JM, Chopineau J, Bazin JE. A pharmacokinetic study of 48-hour sevoflurane inhalation using a disposable delivery system (AnaConDa(R)) in ICU patients. Minerva Anestesiol. 2014 Jun;80(6):655-65. Epub 2013 Nov 13. PMID 24226486
- [Background] Soukup J, Selle A, Wienke A, Steighardt J, Wagner NM, Kellner P. Efficiency and safety of inhalative sedation with sevoflurane in comparison to an intravenous sedation concept with propofol in intensive care patients: study protocol for a randomized controlled trial. Trials. 2012 Aug 10;13:135. doi: 10.1186/1745-6215-13-135. PMID 22883020
- [Background] Strosing KM, Faller S, Gyllenram V, Engelstaedter H, Buerkle H, Spassov S, Hoetzel A. Inhaled Anesthetics Exert Different Protective Properties in a Mouse Model of Ventilator-Induced Lung Injury. Anesth Analg. 2016 Jul;123(1):143-51. doi: 10.1213/ANE.0000000000001296. PMID 27023766
- [Background] Ware LB, Matthay MA. Alveolar fluid clearance is impaired in the majority of patients with acute lung injury and the acute respiratory distress syndrome. Am J Respir Crit Care Med. 2001 May;163(6):1376-83. doi: 10.1164/ajrccm.163.6.2004035. PMID 11371404